CLINICAL TRIAL: NCT03193736
Title: A Prospective, Open, Multicenter Clinical Trial With One Cohort Analysing the Efficacy and Safety of MINIject in Patients With Open Angle Glaucoma Uncontrolled by Topical Hypotensive Medications
Brief Title: MINIject in Patients With Open Angle Glaucoma Uncontrolled by Topical Hypotensive Medications
Acronym: STAR-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: iSTAR Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISM04
Record Dates: First submitted 2017-05-09; First posted 2017-06-21 (Actual); Results first posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- implant (Experimental)
  Interventions: Device: MINIject implant

INTERVENTIONS:
Device: MINIject implant — MINIject implant is used to reduce intra-ocular pressure (IOP) in the eye through a minimally-invasive Glaucoma surgical intervention.
  The intervention is to be performed as stand-alone surgery.

SUMMARY:
The study will evaluate the efficacy and safety of the implant and intra-ocular pressure (IOP) lowering effects with or without glaucoma medications. The procedure will be a stand-alone surgery. Overall, the patient will be asked to perform several examinations up to 24 months after surgery.

The primary efficacy objective of the present study is to show the IOP reduction under medication 6 months after surgery compared to medicated diurnal IOP at screening.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary or secondary open angle glaucoma during screening/baseline visit or earlier.
* Grade 3 (open, 20-35 degrees) or grade 4 (wide open, 35-45 degrees) according to Shaffer Angle Grading System.
* Glaucoma not adequately controlled

Exclusion Criteria:

* Diagnosis of glaucoma other than open angle glaucoma
* Grade 2, grade 1 and grade 0 according to Shaffer Angle Grading System.
* Neovascular glaucoma in the study eye
* Prior glaucoma surgery in the study eye
* Clinically significant corneal disease
* Patients with poor vision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2019-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zubair Hussain, PhD, Study Director — iSTAR Medical
Locations (2):
- Maxivision Eye Hospital, Hyderabad, Telangana, India
- Clinica de ojos Orillac-Calvo, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Denis P, Hirneiss C, Durr GM, Reddy KP, Kamarthy A, Calvo E, Hussain Z, Ahmed IK. Two-year outcomes of the MINIject drainage system for uncontrolled glaucoma from the STAR-I first-in-human trial. Br J Ophthalmol. 2022 Jan;106(1):65-70. doi: 10.1136/bjophthalmol-2020-316888. Epub 2020 Oct 3. PMID 33011690

RESULTS

PARTICIPANT FLOW:
Groups:
- Implant: MINIject implant: MINIject implant is used to reduce intra-ocular pressure in the eye through a minimally-invasive Glaucoma surgical intervention.
  The intervention is to be performed as stand-alone surgery.
Period: Overall Study
Arm/Group | Implant
Started | 26
Received Implant | 25
Completed | 21
Not Completed | 5
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1
Not completed — implant not received | 1

BASELINE CHARACTERISTICS:
Population: 26 patients met eligibility criteria and underwent MINIject implantation surgery. These participants represent safety reporting population.
Arm/Group | Implant
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 9
  Asian | 10
  Caucasian | 0
  Other | 7
Region of Enrollment [Number; unit: participants]
  Panama | 16
  India | 10
primary open-angle glaucoma [Count of Participants; unit: Participants] | 26

OUTCOME MEASURES:

1. Primary Outcome: Change in Medicated Diurnal Intra-ocular Pressure (IOP) at 6 Months Post-implantation
Description: Change of Medicated diurnal IOP [mmHg] from pre-implantation Baseline to 6 months post-implantation, with or without the use of the allowed concomitant glaucoma hypotensive medication
Time Frame: 6 months after implantation surgery
Population: patients who received MINIject implant and were present at both Baseline and 6-month follow-up visit
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Implant
Number analyzed (Participants) | 24
mmHg | -8.95 (3.7)

ADVERSE EVENTS:
Time Frame: 2 years post-implantation
Arm/Group | Implant
All-Cause Mortality (participants affected / at risk) | 2/26
Serious Adverse Events (participants affected / at risk) | 2/26
Other Adverse Events (participants affected / at risk) | 21/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implant (N=26)
death (General disorders) | 1 (1) — death during sleep from unknown cause
pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — pancreatic carcinoma resulting in death
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Implant (N=26)
Anterior Chamber inflammation (Eye disorders) | 8 (8)
Visual acuity reduced (Eye disorders) | 8 (9)
Visual Field Defect (Nervous system disorders) | 7 (7) — >3dB (decibel) worsening from baseline value, even if transient, reported
Intraocular Pressure increased (Investigations) | 5 (6) — *Only one patient had a mean intraocular pressure (IOP) increase, which fulfilled the protocol definition of substantial IOP increase (≥10 mmHg higher than screening IOP after the 1-month postoperative visit).
Lenticular opacities (Eye disorders) | 5 (5)
Hyphaema (Injury, poisoning and procedural complications) | 3 (4)
Conjunctival haemorrhage (Eye disorders) | 2 (2)
eye pain (Eye disorders) | 2 (2)
eye pruritus (Eye disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* first publication to be made by Sponsor as part of publication of results obtained from all sites participating in the study
* intended manuscript to be submitted to Sponsor for review min 60 days in advance, proposals for changes submitted by Sponsor to be taken into consideration by Principal Investigator, unless they interfere with scientific nature or neutrality of the publication
* Sponsor may demand postponement of publication by max 90 days to protect intellectual property rights

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-17): https://cdn.clinicaltrials.gov/large-docs/36/NCT03193736/Prot_SAP_000.pdf